CLINICAL TRIAL: NCT04947007
Title: Comparison of the Efficacy of Different Local Anesthetic Dosage in Suprascapular and Axillary Blocks in Shoulder Arthroscopy Surgeries
Brief Title: Comparison of Different Local Anesthetic Dose in Suprascapular and Axillary Blocks in Shoulder Arthroscopies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020/1830
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative
Keywords: suprascapular nerve block; axillary nerve block; Regional Anesthesia; Analgesic consumption; Postoperative analgesia; Numeric rating scale
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Isotonic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Active Comparator): In this group, US guided suprascapulary and axillary nerve block will be performed with 15cc+15c local anesthetic.
  Interventions: Drug: Bupivacaine hydrogen chloride (HCl) 0.025 % in 15+15 ML Injection
- Group 2 (Active Comparator): In this group, US guided suprascapulary and axillary nerve block will be performed with 10cc+10c local anesthetic.
  Interventions: Drug: Bupivacaine HCl 0.025 % in 10+10 ML Injection
- Group 3 (Active Comparator): In this group, US guided suprascapulary and axillary nerve block will be performed with 5cc+5c local anesthetic.
  Interventions: Drug: Bupivacaine HCl 0.025 % in 5+5 ML Injection
- Group 4 (Active Comparator): In this group, US guided suprascapulary and axillary nerve block will be performed with serum physiologic.
  Interventions: Drug: Isotonic solution

INTERVENTIONS:
Drug: Bupivacaine hydrogen chloride (HCl) 0.025 % in 15+15 ML Injection — In this group, US guided suprascapulary and axillary block will be performed with 15 ml +15 ml 0.025% bupivacaine for each block site using a 22 gauge 10 mm block needle.
  Other Names: Marcaine
  Arms: Group 1
Drug: Bupivacaine HCl 0.025 % in 10+10 ML Injection — In this group, US guided suprascapulary and axillary block will be performed with 10 ml +10 ml 0.025% bupivacaine for each block site using a 22 gauge 10 mm block needle.
  Other Names: Marcaine
  Arms: Group 2
Drug: Bupivacaine HCl 0.025 % in 5+5 ML Injection — In this group, US guided suprascapulary and axillary block will be performed with 5 ml +5 ml 0.025% bupivacaine for each block site using a 22 gauge 10 mm block needle.
  Other Names: Marcaine
  Arms: Group 3
Drug: Isotonic solution — In this group, US guided suprascapulary and axillary block will be performed with isotonic solution
  Other Names: serum physiologic
  Arms: Group 4

SUMMARY:
The research is designed as a single-center, prospective, randomized double-blind study. The patients undergoing shoulder arthroscopy surgery in Istanbul University, Istanbul Faculty of Medicine, Department of Orthopedics and Traumatology will be included. Patients who are legally authorized to make decisions on their behalf will be informed about the research and their written consent will be obtained. Patients who do not give consent will be excluded. Ultrasonography (USG) guided combined suprascapular and axillary block will be performed routinely for postoperative analgesia. After the block is performed, general anesthesia will be applied. The patients will be divided into 4 groups. Three different doses of local anesthetic will be given to patients (30 cc vs 20 cc vs 10 cc). Local anesthetic dose will be the same for suprascapular and axillary blocks. The fourth group will be sham control. Pain score will be determined by visual pain scoring (VAS) and analgesic consumption will be provided by the use of a patient controlled analgesia (PCA) device with intravenous morphine applied in routine practice to all four groups at the postoperative 1, 4, 8,12 and 24 hours. Patient will be observed for postoperative nausea and vomiting, first time to mobilization, length of hospital stay, analgesic consumption and satisfaction of surgeon and patient.

DETAILED DESCRIPTION:
The investigators research was designed as a single-center, prospective, randomized double-blind study.

After the approval of the Ethics Committee, the study will start and is aimed to be completed in 6 months. The patients consecutively undergoing shoulder arthroscopy surgery in Istanbul University Istanbul Faculty of Medicine, Department of Orthopedics and Traumatology will be included. Patients who are legally authorized to make decisions on their behalf will be informed about the research and their written consent will be obtained. Patients who do not give consent will not be included in the study.

Preoperative evaluation of the patients will include detailed history, demographic and clinical parameters including gender, age, indication for shoulder arthroscopy, creatinine, chronic disease history will be recorded. Patients will be taken to the operating room after premedication with 2 mg midazolam and 50 mg fentanyl.

Patients will be monitored for rhythm, blood oxygen and pressure in the operating room. Ultrasonography (USG) guided suprascapular and axillary block will be performed. Suprascapular and axillary block will be done for postoperative analgesia. After the block is done, general anesthesia will be applied. In this study there will be four groups with the control group included. For the first group 15cc+15cc , for the second group 10cc+10cc for the third group 5cc+5cc of local anesthetic will be injected. The fourth group will be sham control.

Pain score will be determined by visual pain scoring (VAS) and analgesic consumption will be provided by the use of a patient controlled analgesia (PCA) device with intravenous morphine applied in routine practice to all four groups at the postoperative 1, 4, 8,12 and 24 hours. Patients will be followed up for 48 hours postoperatively in routine practice. They will be observed for postoperative nausea and vomiting, first mobilisation time, lenght of hospital stay, analgesic consumption and surgent and patient satisfaction.

Before the study, it was determined that at least 132 patients should be collected in the power analysis performed with the help of similar literature data. After collecting the demographic data and morphine consumption data of the patients, statistical analysis will be performed with Statistical Package for the Social Sciences (SPSS). The investigators study does not contain any modifications other than the investigators daily routine practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total shoulder arthroscopy surgery
* Patients with American Society of Anesthesiology (ASA) Class 1-3

Exclusion Criteria:

* Refusal of regional anesthesia
* Infection on the local anesthetic application area
* Patients with known coagulopathy
* Known allergy against local anesthetics
* Anatomical difficulties to perform supra scapular and axillary blocks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (0-10) pain scores for patients | 48 hours
  The VAS (Visual Analog Scale, 0 ''no pain'', to 10, ''the worst pain possible'')

SECONDARY OUTCOMES:
Opioid (mg) consumption | postoperative period up to 48th hours.
  Opioid (mg) consumption

OTHER OUTCOMES:
Time of onset of narcotic analgesic need | postoperative period up to 48th hours.
  (If VAS > 4, morphine 0.05 mg/kg IV will be administered as rescue analgesia additional analgesia and maximum will be increased to 10 mg.
Incidence of side effects | postoperative period up to 48th hour
  Incidence of nausea and vomiting
Time until postoperative first mobilization | Up to 48 hours
  First mobilization time
Length of hospital stay | Through study completion, an average of 1 week
  Hospitalization
Patient satisfaction | postoperative period up to 48th hours and postoperative in the first month
  Satisfaction score; 0- very unsatisfied, 3- very satisfied
Surgeon satisfaction | postoperative period up to 48th hours and postoperative in the first month
  Satisfaction score; 0- very unsatisfied, 3- very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Nil R Kirsan, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Lee JJ, Kim DY, Hwang JT, Song DK, Lee HN, Jang JS, Lee SS, Hwang SM, Moon SH, Shim JH. Dexmedetomidine combined with suprascapular nerve block and axillary nerve block has a synergistic effect on relieving postoperative pain after arthroscopic rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4022-4031. doi: 10.1007/s00167-020-06288-8. Epub 2020 Sep 25. PMID 32975624
- [Background] Ozkan D, Cemaloglu S, Catma FM, Akkaya T. Effects of suprascapular and axillary nerve block on postoperative pain relief sevoflurane consumption and visual clarity in arthroscopic shoulder surgery. Agri. 2020 Jan;32(1):1-7. doi: 10.14744/agri.2019.04875. PMID 32030694
- [Background] Price D. Optimizing the Combined Suprascapular and Axillary Nerve (SSAX) Block. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):122. doi: 10.1097/AAP.0000000000000518. No abstract available. PMID 27997490
- [Background] Marty P, Rontes O, Delbos A. A Comparison of Combined Suprascapular and Axillary Nerve Blocks to Interscalene Block: Interpret With Caution. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):273-274. doi: 10.1097/AAP.0000000000000551. No abstract available. PMID 28207648